CLINICAL TRIAL: NCT06923917
Title: European Registry of Acutely Decompensated Pulmonary Hypertension
Brief Title: European Registry of Acutely Decompensated Pulmonary Arterial Hypertension
Acronym: PHAROS Acute
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Respiratory Society (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250036
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary arterial hypertension; Right heart failure; intensive care; extracorporal life support; transplantation
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with a confirmed diagnosis of pulmonary arterial hypertension managed for acute right hear

SUMMARY:
Acute decompensation of pulmonary hypertension (PH) is associated with a very unfavorable short-term prognosis. However, the development of circulatory support techniques and the possible use of emergency transplantation in recent years has significantly changed the management of patients with refractory right ventricular failure. Nonetheless, there are significant disparities in the management of these patients depending on the organization of the care pathway, the rules for graft allocation, and access to circulatory support across European countries. Moreover, the implementation of these new therapeutic strategies requires the identification of effective prognostic factors and the development of new monitoring techniques. The objective of this collaborative clinical research project is to study the prognostic implications of acute decompensated right heart failure associated with PAH based on a large-scale European multicenter approach using a prospective analysis of clinical, biological, and echocardiographic data.

DETAILED DESCRIPTION:
Precapillary pulmonary hypertension (PH) encompasses a group of diseases characterized by a progressive increase in pulmonary vascular resistance (PVR). The international clinical classification of PH distinguishes these diseases based on their pathophysiological characteristics, clinical presentation, and management. Group 1 [pulmonary arterial hypertension (PAH)] includes diseases characterized by intense remodeling of small pulmonary arteries due to the proliferation of endothelial and smooth muscle cells (1). Within this group, we distinguish isolated pulmonary vascular diseases without comorbidity (idiopathic PAH, "familial" or hereditary PAH, and PAH associated with drug and toxin use) and PAH associated with a concomitant pathology (connective tissue diseases, congenital heart diseases, portal hypertension, HIV infection, schistosomiasis, chronic hemolytic anemias). This distinction is primarily based on the progressive profile of these different conditions. Other forms of precapillary pulmonary hypertension include PH associated with respiratory disease (Group 3), postembolic PH (Group 4), and multifactorial PH (Group 5). Group 2 concerns postcapillary PH, i.e., related to left heart diseases.

Over the past twenty years, PAH has benefited from significant therapeutic innovations resulting from a better understanding of the pathophysiological mechanisms associated with this disease. The currently available treatments primarily target endothelial dysfunction of the pulmonary arteries (2). New therapeutic approaches aiming to reduce pulmonary vascular proliferation in addition to the already available medications are in development. The most advanced therapeutic innovation targets abnormalities related to the receptors of the TGF-ß superfamily (3,4). However, despite the undeniable progress made in the last 20 years, PAH remains an incurable disease that progresses to right ventricular failure and death. The latest epidemiological data from the French PH registry estimate a 25% mortality rate at 3 years (5).

The ability of the right ventricle (RV) to adapt to the progressive increase in PVR is the key prognostic factor for patients with PH (6). The RV's adaptation to excessive afterload begins with concentric myocardial hypertrophy, aiming to normalize the imposed wall stress. Subsequently, the RV dilates in response to increased pressures. The eccentric hypertrophy combined with excessive dilation of the right cavities often reflects a so-called "maladaptive" phenotype. At this stage, severe systolic and diastolic dysfunction of the RV is observed, associated with left ventricular (LV) diastolic dysfunction due to RV/LV interdependence mechanisms. This phenotype corresponds to the final stage of PH, characterized by the onset of NYHA functional class III or IV dyspnea, the appearance of congestive signs, a risk of syncope, and hemodynamically by chronic elevation of right atrial pressures and a decrease in cardiac output. All these clinical, functional, and hemodynamic parameters are closely correlated with a poor prognosis and result from severe impairment of ventriculo-arterial coupling (1).

Patients in the terminal phase of precapillary PH are thus at high risk of developing acute right heart failure, which is predominantly observed in patients with PAH. This clinical situation corresponds to an imbalance of the RV's adaptive phenomena, leading to an acute worsening of symptoms, typically associated with circulatory failure and, in the most severe cases, multiple organ failure. Despite the highly unfavorable prognosis of this clinical situation (7,8), there is currently no precise consensus on the management of these patients. Their care primarily involves identifying and treating any potential triggering factor, optimizing RV preload, and using inotropes if necessary to improve right ventricular performance and stabilize systemic blood pressure. Alongside symptomatic management, the possibility of intensifying specific PH treatment is systematically considered, aiming to reduce RV afterload (9,10).

Despite this management, some patients develop a scenario of refractory right ventricular failure. Therapeutic options for these patients, which were nonexistent 15 years ago, have significantly developed in recent years with circulatory support on one hand, and emergency heart-lung or double-lung transplantation on the other. Since 2006 for heart-lung transplantation and 2007 for double-lung transplantation, the Biomedicine Agency has implemented a "super-urgent" program allowing these patients, in a situation of acute refractory decompensation despite optimal medical treatment, to have priority access to available grafts within the national territory for a renewable period of 8 days. For the most severe patients, veno-arterial extracorporeal membrane oxygenation (ECMO) circulatory support can be implemented while waiting for transplantation. Currently, this procedure is used in about 20% of patients awaiting heart-lung or double-lung transplantation under super-urgent status for PH.

This therapeutic approach has improved the survival of patients hospitalized in intensive care for acute decompensation of pulmonary hypertension and candidates for transplantation (8). It underscores the importance of managing these patients in expert centers capable of offering all possible therapeutic options, whether medical, interventional, or surgical. One of the key points in managing acute right heart failure in PH involves clinical, hemodynamic, and biological monitoring, necessary to evaluate the patient's prognosis, adapt initiated therapies, and decide on emergency transplantation and/or circulatory support in cases of refractory right ventricular failure.

However, there are likely significant disparities in the management of these patients depending on the organization of care pathways, graft allocation rules, and access to circulatory support. The objective of this clinical research collaboration is to study the prognostic implications of decompensated acute right heart failure associated with PAH using a large-scale, multicenter European approach with prospective analysis of clinical, biological, and echocardiographic data.

3.2. Description of the Elements Under Study The study population consists of patients admitted for acute decompensation of PAH requiring treatment with intravenous diuretics, combined with the use of catecholamines if necessary. This study will in no way influence the management of these patients.

Acute decompensation of right ventricular failure will be defined by the worsening of clinical signs of right heart failure within the month preceding hospital admission, requiring:

* the use of i.v. diuretics for ≥ 2 days
* or inotropes
* or vasopressors This cohort study aims to collect clinical, biological, and echocardiographic data from at least 200 patients admitted for an episode of acute decompensation of PAH within multiple European centers belonging to the ERN-Lung network. Information regarding their therapeutic management during hospitalization and their status (alive without transplantation, transplanted, deceased) at 3 months and one year after inclusion will also be collected. This study will enable the analysis of the prognosis of these patients and the identification of prognostic factors based on the collected parameters.

Feasibility and Consistency of the Working Group This project is part of the European clinical research collaboration project PHAROS, supported by the European Respiratory Society (ERS) and closely related to the European Rare Disease Network ERN-Lung.

The investigative centers participating in this study are part of the ERN-Lung network and have already collaborated on this topic, particularly by participating in a survey on the management of acute decompensations of pulmonary hypertension. The results of this survey were presented at the latest European Respiratory Society congress in September 2023 (Savale et al, "Management of acute decompensated pulmonary arterial hypertension: results of the ERS Clinical Research Collaboration PHAROS survey").

Expected Results and Perspectives / Hypotheses / Justification of Public Interest Currently, there are very few studies, primarily retrospective, single-center, and with small sample sizes, that describe the characteristics of patients with acute decompensation of PAH and their prognosis. Recent developments in the management of these patients, especially with the advancement of circulatory support in right ventricular failure and changes in graft allocation rules, necessitate further understanding of the characteristics of these patients and their prognostic parameters.

The goal is to improve the management of these patients and better identify potential candidates for emergency transplantation and/or circulatory support. The European ERN-Lung network provides a unique opportunity to gather data from multiple centers and constitute a cohort large enough to identify prognostic parameters that are relevant for the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established diagnosis of pulmonary arterial hypertension (group 1) according to the 2022 ESC/ERS guidelines.
2. Worsening of clinical signs of right heart failure in the month prior to hospital admission requiring the use of:

   * intravenous diuretic therapy for ≥ 2 days
   * or inotropes
   * or vasopressors

Exclusion Criteria:

1. Patients with non-group 1 pulmonary hypertension
2. Shock due to a cause other than right heart failure
3. Person unable to provide written informed consent (person deprived of liberty by judicial or administrative decision)
4. Person who is the subject of a legal protection measure (tutelage, guardianship, safeguard of justice)
5. Person under psychiatric care
6. Patient's objection to the use of their data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient hospitalized with a confirmed diagnosis of pulmonary arterial hypertension (group 1) according to the latest European guidelines of 2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
3-months mortality/lung transplantation | 3-months post inclusion
  3-months mortality/lung transplantation

SECONDARY OUTCOMES:
12-months mortality/lung transplantation | 12 months most inclusion
  12-months mortality/lung transplantation
Rehospitalization for acute decompensation of PAH within 12 months following inclusion | Within 12 months after inclusion
  Rehospitalization for acute decompensation of PAH within 12 months following inclusion
Proportion of patients treated with catecholamines, placed on ECMO, and transplanted in each center | Within 12 months post inclusion
  Proportion of patients treated with catecholamines, placed on ECMO, and transplanted in each center
Mortality at 3 months following circulatory support | 3 months post inclusion
  Mortality at 3 months following circulatory support
3 and 12-month mortality/lung transplantation in pediatric patients | 3 and 12 months post inclusion
  3 and 12-month mortality/lung transplantation in pediatric patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique hopitaux de Paris, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided